CLINICAL TRIAL: NCT07331233
Title: A Cross-sectional Study on the Impact of Shift Work on Diastolic Dysfunction in Healthcare Workers
Status: Not yet recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202510163RINE
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Diastolic Dysfunction
Keywords: diastolic dysfinction; echocardiography; health worker; shift work

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 60 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- night shift worker: those who need night shift
- day shift workers: those who dont need night shift

SUMMARY:
The goal of this observational cross-sectional study is to assess the prevalence of left ventricular diastolic dysfunction and identify associated risk factors in health-care workers of various ages and both sexes.

The main questions it aims to answer are:

What is the prevalence of diastolic dysfunction among healthcare workers? Which occupational, lifestyle, or clinical factors are associated with abnormal diastolic function in this population?

Researchers will compare health-care workers who dont need night shift with those who have to.

Participants will:

Complete questionnaires regarding demographic information, work schedules, lifestyle factors, and medical history.

Undergo echocardiographic examination to assess diastolic function. Receive basic vital sign by ambulatory blood pressure monotoring.

ELIGIBILITY:
Inclusion Criteria: Healthcare workers at our hospital

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: those who need night work and those who dont
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
diastolic dysfunction | 2026/01~ 2026/12
diastolic dysfunction | from january 2026 to December 2026

IPD SHARING:
Plan to Share IPD: Yes